CLINICAL TRIAL: NCT06657300
Title: Assessment and Comparison of Efficacy of Intra-Articular Platelet Rich Plasma and Corticosteroid on Pain, Hand Function and Pinch Strength in First Carpometacarpal Joint Osteoarthritis Treatment: a Randomized, Prospective, Double-blind Clinical Trial
Brief Title: Assessment and Comparison of Efficacy of Intra-Articular PRP and Corticosteroid in First CMC Joint OA Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AntalyaTRHdabak01
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Thumb Osteoarthritis; Hand Osteoarthritis; Platelet Rich Plasma; Corticosteroid; Intra-articular Injection; Ultrasonography
Keywords: thumb base osteoarthritis; hand osteoarthritis; platelet-rich plasma; corticosteroid; intra-articular injection; ultrasonography
MeSH Terms: interventions — Adrenal Cortex Hormones; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: 10 ml of blood required for PRP preparation was taken from all patients to make the patients blind to which treatment they received. The injectors were taped closed. Outcomes were measured at 1, 3 and 6 months after injection by the physician who performed the initial assessment and was blinded to the type of injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (PRP group) (Experimental): A single dose of 1 ml PRP (Vacusera) was injected into the 1st CMC joint of the first group.
  Interventions: Drug: PRP
- Group 2 (CS group) (Experimental): A single dose of 20 mg of methyl-prednisolone (Depo-Medrol) (complemented to 1 ml by adding 0.5 ml of saline) was injected to the 1st CMC joint of the second group
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: PRP — A single dose of 1 ml PRP (Vacusera) was injected into the 1st CMC joint of the first group. Injection was performed under USG (Clarius; L7 HD Linear Ultrasound Scanner) guidance by the same physician after skin sterilization.
  Other Names: Platelet-rich plasma
  Arms: Group 1 (PRP group)
Drug: Corticosteroid — A single dose of 20 mg(1ml) of methyl-prednisolone (Depo-Medrol) (complemented to 1 ml by adding 0.5 ml of saline) was injected to the 1st CMC joint of the second group. Injection was performed under USG (Clarius; L7 HD Linear Ultrasound Scanner) guidance by the same physician after skin sterilization.
  Other Names: depo-medrol
  Arms: Group 2 (CS group)

SUMMARY:
Aim: We aim to determine and compare the efficiency of single dose intra-articular (IA) platelet rich plasma (PRP) and corticosteroid (CS) injections for the treatment of first carpometacarpal joint osteoarthritis (1. CMC OA) on the basis of pain, hand function and pinch strength.

Material and Method: Sixty patients meeting the criteria were included in the study. Patients were randomized into Group 1 (PRP group) or Group 2 (CS group). Patients were evaluated by Visual Analogue Scale (VAS), Duruoz Hand Index (DHI) and pinch meter for pain and function.

DETAILED DESCRIPTION:
Osteoarthritis(OA) which is the most prevalent form of arthritis, is a degenerative process eroding articular cartilage. Joints affected most commonly include hand, knee, hip and spine.The trapeziometacarpal joint of the thumb (CMC) is a common source of pain due to OA. Age adjusted prevalence of rhizarthrosis is reported as 5-17% in men and 7-21% in women. Although the effect of the CMC osteoarthritis (rhizarthrosis) on hand function and strength have been reported, it is likely underdiagnosed in clinical practice. Conservative treatment modalities range from therapy, orthoses, modification of daily activities to intraarticular injection in early stages. For patients who fail conservative measures or advanced stages, surgical treatment options are indicated.

Platelet-rich plasma (PRP) is the processed fraction of autologous peripheral blood with a platelet concentration above the baseline. PRP therapies have been used in the treatment of dejenerative joint disease and also in different fields of medicine for more than two decades. The rationale underlying the PRP therapy in OA is to stimulate the tissue repair and regeneration via growth factors and bioactive molecules involved in basic pathways such as inflammation, angiogenesis and cell migration in alpha granules of platelets. The studies evaluating the theuropatic effect of PRP in osteoarthritis generally include its application in the knee, hip and shoulder joints. There is very few article reporting the application of PRP in rhizarthrosis.

2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee suggests "no recommendation in regard to osteoarthritis of the hand". Same guideline suggest that " intraarticular glucocorticoid injection is conditionally, rather than strongly, recommended for hand osteoarthritis. In "2018 update of the EULAR recommendation fort he management of hand osteoarthritis" did not mention the PRP application for hand osteoarthritis.

In our prospective, randomised, double-blind, clinical study we aimed to compare the results of the intraarticular application of corticosteroid and PRP in early stages of the rhizarthrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in the first carpometacarpal joint for at least 3 months
2. Patient diagnosed with rhizarthrosis which is classified as stage I-II-III according to Eaton-Littler classification on direct graphy,
3. Patient aged 40-80 years who understood and accepted the written consent

Exclusion Criteria:

1. Patient who has no intraarticular injection in the last 3 months.
2. Oral and/or parenteral corticosteroid usage.
3. Diacerein, chondroitin sulfate, glucosamine sulfate usage.
4. Regular nonsteroidal anti-inflammatory drug usage.
5. Oral anticoagulants and acetylsalicylic acid usage.
6. History of rheumatological, inflammatory, autoimmune or hematological diseases.
7. History of neurological diseases such as cervical radiculopathy, parkinson's disease, stroke or polyneuropathy.
8. History of 1th CMC joint trauma or surgery
9. Shoulder, elbow, wrist tendinopathy or soft tissue disorder in the same extremity and De Quervain's tenosynovitis, Duputyren's contracture or trigger finger.
10. Liver or kidney dysfunction
11. Local or systemic infections
12. Pregnant or lactating patient
13. History of malignancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline , 1st month, 3rd month, 6th month
  The patient's symptoms were filled in, with the VAS score increasing from 0 to 10. The end of a 10 cm line with 0 cm indicating no complaints (best) and the end with 10 cm indicating very severe complaints (worst).

SECONDARY OUTCOMES:
Duruoz Hand Index (DHI) | Baseline , 1st month, 3rd month, 6th month
  DHI score, which quickly evaluates hand problems, consists of 18 questions.
Pinch strength (thumb grip strength) | Baseline , 1st month, 3rd month, 6th month
  Pinch strength was determined by pincmeter (Jamar Digital Pinchmeter). The three types of thumb grip strengths; palmar grip strength, lateral grip strength, and end-to-end grip strength were measured. Each type of pinch measurements was performed 3 times by 1 minute intervals and mean of these three measurements was accepted as end result.

CONTACTS AND LOCATIONS:
Overall Officials: Nimet Ezgi Dabak, M.D., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Muratpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No